CLINICAL TRIAL: NCT02279992
Title: CSMC IIT: Pilot Study of Phosphodiesterase-V Inhibition to Increase Intratumoral Concentration of Carboplatin in Patients With Recurrent High Grade Gliomas and Brain Metastases
Brief Title: Pilot Study of Vardenafil and Carboplatin in Patients With Gliomas and Brain Metastases
Acronym: LevitraCarbo
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Unable to accrue to the study. Original PI no longer with the institute.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSMC IIT: Levitra Carboplatin; Pro00017009 (Other: Cedars-Sinai Medical Center)
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Glioma; Brain Neoplasms; Brain Metastasis
Keywords: Malignant Glioma; Brain Neoplasms, Malignant; Brain metastasis
MeSH Terms: conditions — Glioma; Brain Neoplasms | interventions — Vardenafil Dihydrochloride; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vardenafil + Carboplatin (Experimental): Vardenafil (Levitra®) 20 mg oral administered 1 hour prior to start of craniotomy + Carboplatin (Paraplatin®) 100 mg IV administered over 30 minutes at the start of craniotomy
  Interventions: Drug: Vardenafil; Drug: Carboplatin
- Carboplatin Alone (Active Comparator): Carboplatin (Paraplatin®) 100 mg IV administered over 30 minutes at the start of craniotomy
  Interventions: Drug: Carboplatin

INTERVENTIONS:
Drug: Vardenafil
  Other Names: Levitra®; Phospodiesterase-V Inhibitor
  Arms: Vardenafil + Carboplatin
Drug: Carboplatin
  Other Names: Paraplatin®

SUMMARY:
This is a randomized pilot study to investigate the ability of a phosphodiesterase-V inhibitor (vardenafil) to increase the concentration of systemically delivered chemotherapy, carboplatin, in patients with recurrent malignant gliomas or metastatic brain cancer. This study will also determine the toxicity and tolerability of a phosphodiesterase-V inhibitor (vardenafil) in combination with intravenous carboplatin for patients with recurrent malignant gliomas or metastatic brain cancer.

DETAILED DESCRIPTION:
Twenty patients (10 pts with recurrent malignant glioma and 10 pts with metastatic brain tumor) will be randomly assigned to receive either a phosphodiesterase-V inhibitor (vardenafil) followed by carboplatin or carboplatin alone. All patients will have tumor resection performed from 2 to 6 hours after administration of carboplatin. Using high performance liquid chromatographic (HPLC) or ELISA methodology, carboplatin levels will be determined from both serum and resected tumor tissue. Patients will be followed for four weeks after craniotomy for toxicity associated with the administration of carboplatin and a phosphodiesterase-V inhibitor plus carboplatin.

These data will provide quantitative measures of intratumoral carboplatin levels with and without alteration of blood/tumor barrier (BTB) permeability with vardenafil.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent malignant glioma or metastatic brain cancer requiring craniotomy for gross total resection, subtotal resection or biopsy
* Previously histopathologically proven glioma or radiographic appearance of metastatic lesion with a primary neoplasm that is known to metastasize to the brain
* Patients must have a Karnofsky performance status ≥ 60% (i.e. the patient must be able to care for himself/herself with occasional help from others)
* Patients must have normal hematologic, renal and liver function (i.e. Hemoglobin >10 gm/dl, Absolute neutrophil count ≥ 1500/mm3, Platelets ≥ 100,000/mm3, creatinine ≤ 1.5 mg/dl or Cr Clearance ≥ 60 mL/min, total bilirubin ≤ 1.5 mg/dl, transaminases ≤ 4 times above the upper limits of the institutional normal.
* Patients must be able to provide written informed consent

Exclusion Criteria:

* Patients with serious concurrent infection or medical illness, which would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety
* Patients who are pregnant or breast-feeding
* Patients receiving concurrent therapy for their tumor (i.e. chemotherapeutics or investigational agents)
* Allergy to 5HT-(3) receptor antagonist including tropisetron, ondansetron
* Patients on enzyme-inducing anticonvulsants (Dilantin, Tegretol, Phenobarbital)
* Patients with unstable angina or serious cardiovascular disease
* Known HIV positivity or AIDS-related illness
* History of allergic reaction to platinum compounds or mannitol
* Medical conditions requiring the use of oral nitrates
* Patients on alpha-1 adrenergic blockers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-03-27 (Actual); Primary Completion 2013-10-13 (Actual); Study Completion 2016-02-11 (Actual)

PRIMARY OUTCOMES:
Concentration of intratumoral carboplatin in tumor tissue and serum samples | At the time of tumor resection

SECONDARY OUTCOMES:
Safety and tolerability of vardenafil in combination with carboplatin using common terminology criteria for adverse events (CTCAE) version 3.0 | From baseline to 1 month post-resection

CONTACTS AND LOCATIONS:
Overall Officials: Surasak Phuphanich, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States